CLINICAL TRIAL: NCT06244056
Title: Stellate Ganglion Block as Novel Treatment for Heart Failure Patients
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mina sobhi said fam (Other)
Responsible Party: Sponsor-Investigator, Mina sobhi said fam, resident doctor, Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Stellate Ganglion Block 2023
Record Dates: First submitted 2023-11-17; First posted 2024-02-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Stellate Ganglion Block

STUDY DESIGN:
Intervention Model Description: A stellate ganglion block is performed by a medical professional in a sterile setting. Firstly Position of patient: Semi-lateral decubitus position, with the neck turned contralateral. Using Probe of ultrasound: Linear 6-13 MHz to guide the needle to the stellate ganglion , The skin at the injection site is cleaned with an antiseptic solution to reduce the risk of infection. A local anesthetic is injected into the skin and deeper tissues to numb the area. Needle:25G 1.5 inch or 22G 3.5 inch is inserted through the skin and deeper tissues until it reaches the stellate ganglion.Once the needle is in the correct position, 3-5 mL of local anesthetic (0.25-0.5% bupivacaine) The procedure typically takes about 15-20 minutes.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Narrow QRS complex Heart failure patients (No Intervention): Narrow QRS complex Heart failure patients with optimal medical treatment.
- : Narrow QRS complex Heart failure patients (Active Comparator): : Narrow QRS complex Heart failure patients with optimal medical treatment with stellate ganglion block.
  Interventions: Procedure: Stellate Ganglion Block
- Wide QRS complex heart failure patients (Active Comparator): Wide QRS complex heart failure patients with optimal medical treatment who were non responders to CRT( retrospective and prospective) with stellate ganglion block.
  Interventions: Procedure: Stellate Ganglion Block

INTERVENTIONS:
Procedure: Stellate Ganglion Block — A stellate ganglion block is performed by a medical professional in a sterile setting. Firstly Position of patient: Semi-lateral decubitus position, with the neck turned contralateral. Using Probe of ultrasound: Linear 6-13 MHz to guide the needle to the stellate ganglion , The skin at the injection site is cleaned with an antiseptic solution to reduce the risk of infection. A local anesthetic is injected into the skin and deeper tissues to numb the area. Needle:25G 1.5 inch or 22G 3.5 inch is inserted through the skin and deeper tissues until it reaches the stellate ganglion.Once the needle is in the correct position, 3-5 mL of local anesthetic (0.25-0.5% bupivacaine) The procedure typically takes about 15-20 minutes.
  Arms: : Narrow QRS complex Heart failure patients; Wide QRS complex heart failure patients

SUMMARY:
Stellate Ganglion Block as Novel Treatment for Heart Failure Patients

DETAILED DESCRIPTION:
Stellate Ganglion Block as Novel Treatment for Heart Failure Patients

ELIGIBILITY:
Inclusion Criteria:

* Age 18 : 70 years old.
* NYHA Class III-IV Heart Failure.
* Heart failure with a reduced ejection fraction (HFrEF) LVEF ≤ 40% calculated using 2D echocardiography and Biplane Simpson's .
* Optimal tolerated Medical Therapy for Heart Failure.

Exclusion Criteria:

* Active Malignancy.
* Acute heart failure including pulmonary edema or cardiogenic shock.
* Severe, life-threatening non-cardiac disease.
* Pregnancy.
* Localized infection.
* Coagulopathy or anticoagulated patients.
* Refused this procedure.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2024-02-05 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Change of left ventricular ejection fraction (LVEF). | 3 month
  Change of left ventricular ejection fraction (LVEF).
Change of NYHA classification. | 3 month
  Change of NYHA classification.

SECONDARY OUTCOMES:
Change of 6 minutes walking test. | 3 month
  Change of 6 minutes walking test.
Heart failure hospitalization. | 3 month
  Heart failure hospitalization.
Vascular complications and safety issues. | 3 month
  Vascular complications and safety issues.
Cardiovascular death. | 3 month
  Cardiovascular death.

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Assiut University, Asyut
  - Assiut university, Asyut